CLINICAL TRIAL: NCT03780491
Title: Understanding and Addressing Patient and Provider Preferences Around Discussions of Cost of Breast Cancer Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Cindy Matsen, MD, Assistant Professor, Physician, University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 114421
Record Dates: First submitted 2018-12-17; First posted 2018-12-19 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): The first 50 patients will have usual care with providers conducting the visit in their typical manner.
- Cost Discussion (Experimental): The second group of 50 patients will be the intervention group where the providers will have a discussion of cost emphasizing five points: 1) Cancer care is expensive and it is normal to be concerned about cost. 2) We will recommend treatments for your cancer based on what we think gives you the best chance of doing well, not based on the cost of the treatment. 3) Because of how complex our healthcare system is, it is very hard for your doctors to know what your costs will be, but we will do our best to give you some general information. 4) We have resources available to help you get more specific information so that you can plan appropriately. 5) Do you have any specific concerns about cost that you'd like to share with me?
  Interventions: Other: Cost Discussion

INTERVENTIONS:
Other: Cost Discussion — The second group of 50 patients will be the intervention group where the providers will have a discussion of cost emphasizing five points: 1) Cancer care is expensive and it is normal to be concerned about cost. 2) We will recommend treatments for your cancer based on what we think gives you the best chance of doing well, not based on the cost of the treatment. 3) Because of how complex our healthcare system is, it is very hard for your doctors to know what your costs will be, but we will do our best to give you some general information. 4) We have resources available to help you get more specific information so that you can plan appropriately. 5) Do you have any specific concerns about cost that you'd like to share with me?
  Arms: Cost Discussion

SUMMARY:
The investigators hypothesize that many cancer patients desire discussions of cost as part of their care, but that preferences for having cost discussions with their physicians vary. Further, the investigators hypothesize that providers can introduce the topic of cost into clinical conversations in a balanced way and that this will improve shared decision making and patient uptake of offers of financial counseling which will lead to improved financial well-being, patient satisfaction with providers, and satisfaction with treatment decisions.

Aim 1: Further understand patient preferences and attendant associations for cost discussions through a patient survey of newly diagnosed breast cancer patients.

Aim 2: Study the influence of provider communication about cost on shared decision making, uptake of financial counseling, financial well-being and satisfaction through an intervention to encourage discussion of cost by breast cancer surgeons with subsequent referral to financial counseling.

DETAILED DESCRIPTION:
Newly diagnosed breast cancer patients over the age of 18 will be eligible for participation. All stages of disease will be included. Eligible participants will be approached in clinic. Those interested will provide written, informed consent at the time of their clinic visit. All participants will be asked to complete baseline surveys consisting of the InCharge Financial Distress/Financial Well Being scale (IFDFW),[24] the Maximizer-Minimizer Scale,[25] and a three question, 5-point Likert scale survey about desire for cost information (1: How concerned are participants about the cost of their cancer care? 2: How interested are participants in discussing cost of care with their doctors? 3: How interested are participants in meeting with a financial counselor about the costs of their care?) Demographic information including age, race and ethnicity, marital status, number of children, current employment status of self and spouse, and education level will be included. To decrease participant burden and encourage study participation, only the three question survey will be required to be completed prior to the visit. The other survey components (IFDFW and Max-Min Scale) can be completed after the visit, but prior to seeing a financial counselor. Participants will be offered a $10 giftcard of their choice (grocery store, Starbucks, Amazon, or gas) at each survey timepoint ($20 total) for participation.

For this study, the investigators will use a pre and post design with 100 total participants. All visits will be audiorecorded, transcribed, and coded for whether cost was discussed in the control group and whether the intervention was successfully implemented in the intervention group as well as shared decision making using the observer-OPTION scale. The first 50 patients will have usual care with providers conducting the visit in their typical manner.

From our past studies, study team discusses cost in 15% of visits, though these discussion tend to be very superficial. The second group of 50 patients will be the intervention group where the providers will have a discussion of cost emphasizing five points: 1) Cancer care is expensive and it is normal to be concerned about cost. 2) The investigators will recommend treatments for the participants' cancer based on what the investigators think gives them the best chance of doing well, not based on the cost of the treatment. 3) Because of how complex our healthcare system is, it is very hard for their doctors to know what their costs will be, but the investigators will do our best to give participants some general information. 4) The investigators have resources available to help participants get more specific information so that participants can plan appropriately. 5) Do participants have any specific concerns about cost that participants would like to share with me? The investigators will encourage study team to have this discussion at the beginning of the consult, but the exact timing will be according to study team judgment.

After the visit, all patients will complete a patient satisfaction survey and will be offered a referral to a financial counselor at our institution. Financial counseling will take place per our usual institutional protocols either in person or over the phone. Our financial counselors are aware that they may see an increased volume of patients during the study period and the investigators will provide funding to cover the increased need. Volume will be tracked during the study period and compared to the non-study period and between the groups.

At the first three to six-month follow-up visit with the surgeon, participants will again complete the IFDFW, a validated patient satisfaction scale[26], and the Satisfaction with Decision Scale.[27].

Data will have personal health identifiers removed from the data for the analysis portion of the study. PHI will not be reused without first seeking IRB approval.

The investigators will enroll 100 patients in two consecutive groups of 50. This gives us 80% power with a two sided significance level of 0.05 for seeing a 27-30% improvement (0.27-0.3 higher score) in our primary outcome of financial well-being as measured by the IFDFW in the intervention group at 3-6 months after the initial visit; the average pre-score on the IFDFW is 5.52 in past studies with improvements of 0.32-1.18 seen in past studies of education interventions to improve financial well-being.[24] This level of difference may not be achievable with this small study, but will provide data for powering a larger study.

Maximizer-Minimizer status, uptake of financial counseling, patient satisfaction, decision satisfaction, and demographic variables will be evaluated for associations with financial well-being using logistic regression methods.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* All patients who present to Huntsman Cancer Hospital/University of Utah for a newly diagnosed breast cancer surgical consultation.

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-11-05 (Actual); Primary Completion 2020-11-16 (Actual); Study Completion 2020-11-16 (Actual)

PRIMARY OUTCOMES:
InCharge Financial Distress/Financial Well-being Scale | 3-6 months after visit
  The InCharge Financial Distress/Financial Well Being scale, an eight-item self-report subjective measure of financial distress/financial well-being. Sores are numeric 1-10. Higher scores indicate higher financial well-being.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

REFERENCES:
- [Background] Altomare I, Irwin B, Zafar SY, Houck K, Maloney B, Greenup R, Peppercorn J. Physician Experience and Attitudes Toward Addressing the Cost of Cancer Care. J Oncol Pract. 2016 Mar;12(3):e281-8, 247-8. doi: 10.1200/JOP.2015.007401. Epub 2016 Feb 16. PMID 26883407
- [Background] Shih YT, Chien CR. A review of cost communication in oncology: Patient attitude, provider acceptance, and outcome assessment. Cancer. 2017 May 15;123(6):928-939. doi: 10.1002/cncr.30423. Epub 2016 Nov 28. PMID 27893929
- [Background] Farina KL. The economics of cancer care in the United States. Am J Manag Care. 2012 Feb;18(1 Spec No.):SP38-9. No abstract available. PMID 22468873
- [Background] Bullock AJ, Hofstatter EW, Yushak ML, Buss MK. Understanding patients' attitudes toward communication about the cost of cancer care. J Oncol Pract. 2012 Jul;8(4):e50-8. doi: 10.1200/JOP.2011.000418. Epub 2012 Feb 28. PMID 23180999
- [Background] Irwin B, Kimmick G, Altomare I, Marcom PK, Houck K, Zafar SY, Peppercorn J. Patient experience and attitudes toward addressing the cost of breast cancer care. Oncologist. 2014 Nov;19(11):1135-40. doi: 10.1634/theoncologist.2014-0117. Epub 2014 Oct 1. PMID 25273078
- [Background] Kelly RJ, Forde PM, Elnahal SM, Forastiere AA, Rosner GL, Smith TJ. Patients and Physicians Can Discuss Costs of Cancer Treatment in the Clinic. J Oncol Pract. 2015 Jul;11(4):308-12. doi: 10.1200/JOP.2015.003780. Epub 2015 May 26. PMID 26015459
- [Background] Hunter WG, Zafar SY, Hesson A, Davis JK, Kirby C, Barnett JA, Ubel PA. Discussing Health Care Expenses in the Oncology Clinic: Analysis of Cost Conversations in Outpatient Encounters. J Oncol Pract. 2017 Nov;13(11):e944-e956. doi: 10.1200/JOP.2017.022855. Epub 2017 Aug 23. PMID 28834684
- [Background] Hunter WG, Zhang CZ, Hesson A, Davis JK, Kirby C, Williamson LD, Barnett JA, Ubel PA. What Strategies Do Physicians and Patients Discuss to Reduce Out-of-Pocket Costs? Analysis of Cost-Saving Strategies in 1,755 Outpatient Clinic Visits. Med Decis Making. 2016 Oct;36(7):900-10. doi: 10.1177/0272989X15626384. Epub 2016 Jan 19. PMID 26785714
- [Background] Alexander GC, Casalino LP, Tseng CW, McFadden D, Meltzer DO. Barriers to patient-physician communication about out-of-pocket costs. J Gen Intern Med. 2004 Aug;19(8):856-60. doi: 10.1111/j.1525-1497.2004.30249.x. PMID 15242471
- [Background] Meropol NJ, Schrag D, Smith TJ, Mulvey TM, Langdon RM Jr, Blum D, Ubel PA, Schnipper LE; American Society of Clinical Oncology. American Society of Clinical Oncology guidance statement: the cost of cancer care. J Clin Oncol. 2009 Aug 10;27(23):3868-74. doi: 10.1200/JCO.2009.23.1183. Epub 2009 Jul 6. PMID 19581533
- [Background] Henrikson NB, Tuzzio L, Loggers ET, Miyoshi J, Buist DS. Patient and oncologist discussions about cancer care costs. Support Care Cancer. 2014 Apr;22(4):961-7. doi: 10.1007/s00520-013-2050-x. Epub 2013 Nov 26. PMID 24276955
- [Background] Bestvina CM, Zullig LL, Rushing C, Chino F, Samsa GP, Altomare I, Tulsky J, Ubel P, Schrag D, Nicolla J, Abernethy AP, Peppercorn J, Zafar SY. Patient-oncologist cost communication, financial distress, and medication adherence. J Oncol Pract. 2014 May;10(3):162-7. doi: 10.1200/JOP.2014.001406. PMID 24839274
- [Background] Jagsi R, Sulmasy DP, Moy B. Value of cancer care: ethical considerations for the practicing oncologist. Am Soc Clin Oncol Educ Book. 2014:e146-9. doi: 10.14694/EdBook_AM.2014.34.e146. PMID 24857095
- [Background] Bakshi, N., et al., Shared decision making or physician advocate for a particular treatment option: A spectrum of approaches to decision making about disease modifying therapies in sickle cell disease. Blood, 2016. 128(22).
- [Background] Makoul G, Clayman ML. An integrative model of shared decision making in medical encounters. Patient Educ Couns. 2006 Mar;60(3):301-12. doi: 10.1016/j.pec.2005.06.010. Epub 2005 Jul 26. PMID 16051459
- [Background] Elwyn G, Cochran N, Pignone M. Shared Decision Making-The Importance of Diagnosing Preferences. JAMA Intern Med. 2017 Sep 1;177(9):1239-1240. doi: 10.1001/jamainternmed.2017.1923. No abstract available. PMID 28692733
- [Background] Elwyn G, Frosch D, Thomson R, Joseph-Williams N, Lloyd A, Kinnersley P, Cording E, Tomson D, Dodd C, Rollnick S, Edwards A, Barry M. Shared decision making: a model for clinical practice. J Gen Intern Med. 2012 Oct;27(10):1361-7. doi: 10.1007/s11606-012-2077-6. Epub 2012 May 23. PMID 22618581
- [Background] Cassel CK, Guest JA. Choosing wisely: helping physicians and patients make smart decisions about their care. JAMA. 2012 May 2;307(17):1801-2. doi: 10.1001/jama.2012.476. Epub 2012 Apr 4. No abstract available. PMID 22492759
- [Background] Janz NK, Wren PA, Copeland LA, Lowery JC, Goldfarb SL, Wilkins EG. Patient-physician concordance: preferences, perceptions, and factors influencing the breast cancer surgical decision. J Clin Oncol. 2004 Aug 1;22(15):3091-8. doi: 10.1200/JCO.2004.09.069. PMID 15284259
- [Background] Jagsi R, Li Y, Morrow M, Janz N, Alderman A, Graff J, Hamilton A, Katz S, Hawley S. Patient-reported Quality of Life and Satisfaction With Cosmetic Outcomes After Breast Conservation and Mastectomy With and Without Reconstruction: Results of a Survey of Breast Cancer Survivors. Ann Surg. 2015 Jun;261(6):1198-206. doi: 10.1097/SLA.0000000000000908. PMID 25654742
- [Background] Altschuler A, Nekhlyudov L, Rolnick SJ, Greene SM, Elmore JG, West CN, Herrinton LJ, Harris EL, Fletcher SW, Emmons KM, Geiger AM. Positive, negative, and disparate--women's differing long-term psychosocial experiences of bilateral or contralateral prophylactic mastectomy. Breast J. 2008 Jan-Feb;14(1):25-32. doi: 10.1111/j.1524-4741.2007.00521.x. PMID 18186862
- [Background] Bhutiani N, Mercer MK, Bachman KC, Heidrich SR, Martin RCG 2nd, Scoggins CR, McMasters KM, Ajkay N. Evaluating the Effect of Margin Consensus Guideline Publication on Operative Patterns and Financial Impact of Breast Cancer Operation. J Am Coll Surg. 2018 Jul;227(1):6-11. doi: 10.1016/j.jamcollsurg.2018.01.050. Epub 2018 Feb 9. PMID 29428232
- [Background] Herrick NL, Unkart JT, Reid CM, Li SS, Wallace AM. Process of Care in Breast Reconstruction and the Impact of a Dual-Trained Surgeon. Ann Plast Surg. 2018 May;80(5S Suppl 5):S288-S291. doi: 10.1097/SAP.0000000000001385. PMID 29489535
- [Background] Meeker CR, Wong YN, Egleston BL, Hall MJ, Plimack ER, Martin LP, von Mehren M, Lewis BR, Geynisman DM. Distress and Financial Distress in Adults With Cancer: An Age-Based Analysis. J Natl Compr Canc Netw. 2017 Oct;15(10):1224-1233. doi: 10.6004/jnccn.2017.0161. PMID 28982748
- [Background] Scherer LD, Caverly TJ, Burke J, Zikmund-Fisher BJ, Kullgren JT, Steinley D, McCarthy DM, Roney M, Fagerlin A. Development of the Medical Maximizer-Minimizer Scale. Health Psychol. 2016 Nov;35(11):1276-1287. doi: 10.1037/hea0000417. Epub 2016 Sep 12. PMID 27617512
- [Background] Presson AP, Zhang C, Abtahi AM, Kean J, Hung M, Tyser AR. Psychometric properties of the Press Ganey(R) Outpatient Medical Practice Survey. Health Qual Life Outcomes. 2017 Feb 10;15(1):32. doi: 10.1186/s12955-017-0610-3. PMID 28183312
- [Background] Holmes-Rovner M, Kroll J, Schmitt N, Rovner DR, Breer ML, Rothert ML, Padonu G, Talarczyk G. Patient satisfaction with health care decisions: the satisfaction with decision scale. Med Decis Making. 1996 Jan-Mar;16(1):58-64. doi: 10.1177/0272989X9601600114. PMID 8717600